CLINICAL TRIAL: NCT03340805
Title: Pragmatic Pediatric Trial of Balanced Versus Normal Saline Fluid in Sepsis: A Pilot Feasibility Study
Acronym: PRoMPT BOLUS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Utah (Other); University of Pennsylvania (Other); University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17-013936
Record Dates: First submitted 2017-11-02; First posted 2017-11-14 (Actual); Results first posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-06

CONDITIONS: Shock, Septic
Keywords: Sepsis; Septic shock; Pediatric; Fluid resuscitation; Saline; Lactated Ringer's; Crystalloid; Mortality; Pragmatic trial; Feasibility
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Ringer's Lactate; Saline Solution

STUDY DESIGN:
Intervention Model Description: Single-center, open-label, randomized pragmatic clinical trial
Masking Description: Study participants, care provider, investigator, and outcomes assessor will not be masked to intervention allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lactated Ringer's fluid (LR) (Experimental): Lactated Ringer's (LR) fluid will be administered to patients randomized to the experimental arm. LR will be used for all fluid boluses and maintenance fluids (supplemental electrolytes are allowed) from time immediately after randomization through 11:59 pm of the next calender day. The determination of when to give fluid, how much fluid to give, how fast to give fluid, and what access to use to administer fluid will remain at the discretion of the treating team.
  Interventions: Drug: Lactated Ringer
- 0.9% "normal" saline fluid (NS) (Active Comparator): 0.9% "normal" saline (NS) fluid will be administered to patients randomized to the active comparator (control) arm. NS will be used for all fluid boluses and maintenance fluids (supplemental electrolytes are allowed) from time immediately after randomization through 11:59 pm of the next calender day. The determination of when to give fluid, how much fluid to give, how fast to give fluid, and what access to use to administer fluid will remain at the discretion of the treating team.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Lactated Ringer — LR is a sterile, nonpyrogenic "balanced" solution used for fluid and electrolyte replenishment via intravenous or intraosseous administration. Each 100 mL of LR contains 600 mg sodium chloride (NaCl), 310 mg of sodium lactate (C3H5NaO3), 30 mg of potassium chloride (KCl), and 20 mg of calcium chloride (CaCl2 · 2H20) with an approximate potential of hydrogen (pH) of 6.5 (6.0 to 7.5).
  Other Names: LR
  Arms: Lactated Ringer's fluid (LR)
Drug: Normal saline — Normal saline solution is an "unbalanced" crystalloid solution containing 154 mEq/L of sodium and 154 milliequivalent (mEq/L) of chloride.
  Other Names: 0.9% Saline; NS
  Arms: 0.9% "normal" saline fluid (NS)

SUMMARY:
The objective of this pilot study is to assess overall feasibility prior to embarking on a larger randomized pragmatic trial comparing the clinical effectiveness of fluid resuscitation with NS versus LR for pediatric patients with suspected septic shock. Necessary feasibility assessments include ensuring appropriate compliance with study fluid in each of the two arms, effectiveness of study enrollment using a pragmatic study design embedded within routine clinical practice, and acceptability of using Exception from Informed Consent (EFIC).

DETAILED DESCRIPTION:
Approximately 5,000 children die from septic shock each year in the US and thousands more die worldwide. Despite widespread implementation of resuscitation protocols, contemporary studies still report 2-6% mortality for children with septic shock treated in the pediatric emergency department (ED). In the investigators' recent survey of the Pediatric Emergency Care Applied Research Network (PECARN), 45% of physicians had treated a child for septic shock in the ED who subsequently died in the hospital in the past two years.

Fluid resuscitation is the cornerstone of resuscitation for hypovolemia and shock, and intravenous fluids are among the most commonly used therapies worldwide. Yet, there remains uncertainty as to the most appropriate fluid type to restore effective blood volume and optimize organ perfusion. In the absence of a clear role for the early use colloids, administration of crystalloid fluids is generally preferred (except in cases of hemorrhage). For septic shock, in particular, crystalloid fluids have long been the standard resuscitative fluid. Crystalloid fluids can be categorized as non-buffered (most commonly 0.9% normal saline [NS]) or buffered/balanced (in the US, this is most commonly lactated Ringer's [LR]) solutions. NS and LR are inexpensive, stable at room temperature, and nearly universally available with identical storage volumes and dosing strategies. Notably, both are also of proven clinical benefit in septic shock and have extensive clinical experience for use in fluid resuscitation of critically ill patients. However, while NS is currently used in 80-95% of cases of septic shock, an increasing body of data now suggest that LR resuscitation may have superior efficacy and safety. Buffered crystalloids, including LR, have demonstrated a 1-4% absolute mortality reduction and up to a 50% lower odds of dialysis compared to NS in observational and non-randomized interventional studies in adult sepsis. Nevertheless, because definitive conclusions have not been able to be drawn from existing observational and non-randomized studies, NS overwhelmingly remains the most commonly used fluid based on historical precedent while controversy remains.

To definitively test the comparative effectiveness of NS and LR, a well-powered randomized controlled trial (RCT) is necessary. A large pragmatic randomized trial embedded within everyday clinical practice provides a cost-efficient and generalizable approach to inform clinicians about best comparative effectiveness of common therapies. Unlike explanatory RCTs, pragmatic trials need heterogeneity in patients, non-study therapies, and settings. To accomplish this, these trials must be large enough to detect small effects and simple enough to incorporate into routine clinical practice. The characteristics of LR and NS provide the ideal scenario for a large pragmatic trial.18 An ED-based trial is necessary to enroll patients at initiation of resuscitation. While any benefit is expected to be small, even a 1-2% absolute reduction in mortality that is in line with prior adult studies would be a clinically important difference by saving the lives of 50-100 children in the US (and many more worldwide) each year. This overall public health impact is commensurate with changing from NS to LR because such a practice change is a simple, cost-neutral shift from largely using NS to largely using LR.

However, before embarking on a large, pragmatic randomized trial that will determine the comparative effectiveness and safety of NS and LR, several concerns regarding feasibility of such a trial need to be addressed including a) ensuring adequate compliance with study fluid administration within each randomized arm using the proposed pragmatic study design, b) determining that a sufficient proportion of patients can be enrolled using the proposed pragmatic study design that will be embedded within routine clinical practice rather than use of a dedicated study team, and c) demonstrating that the study can feasibly be performed using EFIC when enrolling critically ill infants, children, and adolescents into this clinical trial. Demonstrating these feasibility criteria at a single site will strongly support success in a larger, multicenter study that will enroll several thousand patients across the 18 sites comprising Pediatric Emergency Care Applied Research Network (PECARN) to test morbidity and mortality outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age >6 months to <18 years
2. Clinician concern for septic shock, operationalized as:

   1. a "positive" ED sepsis alert confirmed at the physician-led "sepsis huddle" OR
   2. a physician diagnosis of suspected septic shock requiring parenteral antibiotics and fluid resuscitation as per the ED sepsis management pathway
3. administration of at least 20 mL/kg IV/ intraosseous (IO) fluid resuscitation
4. Receipt of ≤40 mL/kg IV/IO crystalloid fluid prior to randomization
5. Additional fluid deemed likely to be necessary to treat poor perfusion, defined as either hypotension or abnormal (either "flash" or >2 second) capillary refill (as determined by clinician's judgment)10
6. Parental/guardian permission (informed consent) if time permits; otherwise, EFIC criteria met

Exclusion Criteria:

1. Clinician judgement that patient's condition deems it unsafe to administer either NS or LR (since patients will be equally likely to receive NS or LR at time of study enrollment), including (but not limited to):

   1. Clinical suspicion for impending brain herniation based on data available at or before patient meets criteria for study enrollment
   2. Known hyperkalemia, defined as non-hemolyzed whole blood or plasma/serum potassium > 6 mEq/L, based on data available at or before patient meets criteria for study enrollment
   3. Known hypercalcemia, defined as plasma/serum total calcium >12 mg/dL or whole blood ionized calcium > 1.35 mmol/L, based on data available at or before patient meets criteria for study enrollment
   4. Known acute fulminant hepatic failure, defined as plasma/serum alanine aminotransferase (ALT) >10,000 U/L or total bilirubin >12.0 mg/dL, based on data available at or before patient meets criteria for study enrollment
   5. Known history of severe hepatic impairment, defined as diagnosis of cirrhosis, "liver failure", or active listing for liver transplant
   6. Known history of severe renal impairment, defined as current dependency on peritoneal dialysis or hemodialysis
   7. Known metabolic disorder, inborn error of metabolism, or primary mineralcorticoid deficiency (e.g., mitochondrial disorder, urea cycle disorder, amino acidemia, fatty acid oxidation disorder, glycogen storage disorder, congenital adrenal hypoplasia, Addison's disease) as reported by subject, LAR or accompanying caregiver, or as listed in the medical record
2. Known pregnancy determined by routine clinical history disclosed by patient and/or legally authorized representative (LAR) (or other accompanying acquaintance)
3. Known prisoner as determined by routine social history disclosed by patient and/or LAR (or other accompanying acquaintance)
4. Known allergy to either normal saline or lactated Ringer's as determined by routine allergy history disclosed by patient and/or LAR (or other accompanying acquaintance) or as indicated in the medical record
5. Indication of prior declined consent to participate based on presence of "PRoMPT BOLUS Opt-Out" bracelet

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2019-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fran Balamuth, MD PhD MSCE, Principal Investigator — Attending Physician, Emergency Department
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weiss SL, Keele L, Balamuth F, Vendetti N, Ross R, Fitzgerald JC, Gerber JS. Crystalloid Fluid Choice and Clinical Outcomes in Pediatric Sepsis: A Matched Retrospective Cohort Study. J Pediatr. 2017 Mar;182:304-310.e10. doi: 10.1016/j.jpeds.2016.11.075. Epub 2017 Jan 4. PMID 28063688
- [Background] Emrath ET, Fortenberry JD, Travers C, McCracken CE, Hebbar KB. Resuscitation With Balanced Fluids Is Associated With Improved Survival in Pediatric Severe Sepsis. Crit Care Med. 2017 Jul;45(7):1177-1183. doi: 10.1097/CCM.0000000000002365. PMID 28437373
- [Background] Semler MW, Rice TW. Saline Is Not the First Choice for Crystalloid Resuscitation Fluids. Crit Care Med. 2016 Aug;44(8):1541-4. doi: 10.1097/CCM.0000000000001941. No abstract available. PMID 27428117
- [Background] Young P. Saline Is the Solution for Crystalloid Resuscitation. Crit Care Med. 2016 Aug;44(8):1538-40. doi: 10.1097/CCM.0000000000001844. No abstract available. PMID 27153047
- See also: PRoMPT BOLUS Website — https://promptbolus.research.chop.edu/
- See also: Children's Hospital of Philadelphia Pediatric Sepsis Program Website — http://www.chop.edu/sepsis

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lactated Ringer's Fluid (LR) | 0.9% "Normal" Saline Fluid (NS)
Started | 24 | 26
Completed | 24 (1 subject withdrew early from study fluid administration but stayed in trial for outcome assessment) | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lactated Ringer's Fluid (LR) | 0.9% "Normal" Saline Fluid (NS) | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24 | 26 | 50
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 3.8 [2.0 to 10.4] | 9.7 [2.6 to 16.3] | 5.8 [2.1 to 12.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 13 | 14 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Non-Hispanic White | 11 | 11 | 22
  Race/Ethnicity: Non-Hispanic Black | 3 | 4 | 7
  Race/Ethnicity: Hispanic | 10 | 9 | 19
  Race/Ethnicity: Asian | 0 | 1 | 1
  Race/Ethnicity: Unknown/Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 24 | 26 | 50
Comorbid Conditions [Number; unit: participants]
  Cancer | 4 | 5 | 9
  Kidney disease | 2 | 1 | 3
  Neurologic dysfunction | 7 | 5 | 12
  Chronic ventilator dependence | 6 | 5 | 11
  Bone marrow or solid organ transplant | 3 | 2 | 5
  Sickle cell disease | 0 | 2 | 2
  Indwelling central venous catheter | 6 | 4 | 10
  Any comorbid condition | 16 | 16 | 32
Site of Infection [Number; unit: participants]
  Bacteremia | 2 | 4 | 6
  Pneumonia/lung infection | 5 | 5 | 10
  Abdominal infection | 1 | 0 | 1
  Urinary Tract Infection | 4 | 3 | 7
  CNS infection | 2 | 3 | 5
  Skin/soft tissue infection | 2 | 3 | 5
  Other | 6 | 6 | 12
  Unknown | 3 | 4 | 7
  Alternative diagnosis other than infection | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Compliance With Study Fluid Administration in the Assigned Study Arm
Description: Proportion of total crystalloids administered as saline in each arm during the intervention phase
Time Frame: up 48 hours after randomization
Measure: Median (Inter-Quartile Range); unit: Proportion of total crystalloids adminis
Arm/Group | Lactated Ringer's Fluid (LR) | 0.9% "Normal" Saline Fluid (NS)
Number analyzed (Participants) | 24 | 26
Proportion of total crystalloids adminis | 0 [0 to 0] | 100 [100 to 100]

2. Secondary Outcome: Enrollment of Eligible Patients
Description: Proportion of eligible patients treated in the pediatric ED who are enrolled, randomized, and treated with study fluid
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Groups:
- All Eligible Patients: All patients age >6 mos to <18 years with clinician suspicion of septic shock who did not meet exclusion criteria
Arm/Group | All Eligible Patients
Number analyzed (Participants) | 59
Participants | 50

3. Secondary Outcome: Acceptability of Enrollment Using "Exception From Informed Consent"
Description: Proportion of eligible patients who meet criteria for EFIC who are enrolled, randomized, and treated with study fluid and do not withdraw prior to completion of the follow-up phase
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Subjects Enrolled Under Exception From Informed Consent: Eligible subjects enrolled under "exception from informed consent" process
Arm/Group | Subjects Enrolled Under Exception From Informed Consent
Number analyzed (Participants) | 44
Participants | 43

4. Other Pre Specified Outcome: Mortality
Description: Proportion of enrolled patients who do not survive
Time Frame: up to 90 days following randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Lactated Ringer's Fluid (LR) | 0.9% "Normal" Saline Fluid (NS)
Number analyzed (Participants) | 24 | 26
Participants | 0 | 1

5. Other Pre Specified Outcome: Hospital-free Days
Description: The number of calendar days alive and out of the hospital between randomization (day 0) and day 27 with death prior hospital discharge defined as "zero" hospital-free days
Time Frame: up to 28 days following randomization
Measure: Median (Inter-Quartile Range); unit: days alive and free of hospitalization
Arm/Group | Lactated Ringer's Fluid (LR) | 0.9% "Normal" Saline Fluid (NS)
Number analyzed (Participants) | 24 | 26
days alive and free of hospitalization | 23 [20 to 25] | 25 [20 to 26]

6. Other Pre Specified Outcome: New Inpatient Dialysis
Description: Proportion treated with any replacement therapy that was not a continuation of pre-hospital chronic therapy
Time Frame: Up to 90 days following randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Lactated Ringer's Fluid (LR) | 0.9% "Normal" Saline Fluid (NS)
Number analyzed (Participants) | 24 | 26
Participants | 0 | 0

7. Other Pre Specified Outcome: Hospital Length of Stay
Description: Measured as the number of calendar days between ED arrival and ED or hospital discharge (whichever occurs later)
Time Frame: up to 90 days following randomization
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Lactated Ringer's Fluid (LR) | 0.9% "Normal" Saline Fluid (NS)
Number analyzed (Participants) | 24 | 26
days | 5 [3 to 8] | 3 [2 to 9]

8. Other Pre Specified Outcome: Adverse Events
Description: Hyperlactatemia, hyperkalemia, hypercalcemia, hypernatremia, hyponatremia, hyperchloremia, therapy for brain herniation
Time Frame: up to four days post-randomization
Measure: Number; unit: adverse events
Arm/Group | Lactated Ringer's Fluid (LR) | 0.9% "Normal" Saline Fluid (NS)
Number analyzed (Participants) | 24 | 26
adverse events | 7 | 18

9. Other Pre Specified Outcome: Adverse Events
Description: Venous thromboembolism
Time Frame: up to seven days post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Lactated Ringer's Fluid (LR) | 0.9% "Normal" Saline Fluid (NS)
Number analyzed (Participants) | 24 | 26
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 7 days
Description: Selective AEs recorded were: Death, Cardiac arrest, Arrhythmia requiring intervention, Vasoactive infusion, ECMO, Invasive mechanical ventilation, Non-invasive mechanical ventilation, Dialysis (not pre-existing), Liver dysfunction, Limb necrosis, Brain herniation, Seizure, Pulmonary embolus, Deep venous thrombosis, Central venous line clot requiring pharmacologic therapy, Bleeding, Hospital infection, Pressure ulcer, IV infiltrate (grade 3 or 4), Rash, and electrolyte abnormalities
Arm/Group | Lactated Ringer's Fluid (LR) | 0.9% "Normal" Saline Fluid (NS)
All-Cause Mortality (participants affected / at risk) | 0/24 | 1/26
Serious Adverse Events (participants affected / at risk) | 4/24 | 2/26
Other Adverse Events (participants affected / at risk) | 11/24 | 12/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lactated Ringer's Fluid (LR) (N=24) | 0.9% "Normal" Saline Fluid (NS) (N=26)
Shock (Cardiac disorders) | 2 (2) | 2 (2) — Requiring vasoactive medications
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) — Requiring invasive ventilation
Death (General disorders) | 0 (0) | 1 (1)
Cerebral edema (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lactated Ringer's Fluid (LR) (N=24) | 0.9% "Normal" Saline Fluid (NS) (N=26)
Hyperlactatemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4) — Hyperlacatatemia > 4 mmol/L
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) — Hyperkalemia >6 mEq/L
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) — Hypercalcemia (ionized calcium > 1.35 mEq/L or total calcium > 12 mEq/L)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) — Hypernatremia >155 mEq/L
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) — Hyponatremia <128 mEq/L
Hyperchloremia (Metabolism and nutrition disorders) | 3 (3) | 7 (7) — Hyperchloremia >110 mEq/L
Thrombosis (Vascular disorders) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (6) — Non-invasive mechanical ventilation
Seizure (Nervous system disorders) | 1 (1) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4)
Liver dysfunction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pressure injury (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/05/NCT03340805/Prot_SAP_000.pdf